CLINICAL TRIAL: NCT01492140
Title: A Randomized, Evaluator-Blind, Bilateral Comparison of an Injection Assistance Device Versus Manual Injections for Delivery of Dermal Fillers in Patients Seeking Aesthetic Correction of the Nasolabial Folds
Brief Title: Injection Assistance Device Versus Manual Injections for Delivery of Dermal Fillers
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: TKL Research, Inc. (Industry)
Collaborators: Nordson Micromedics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NM-11-01
Record Dates: First submitted 2011-12-07; First posted 2011-12-14 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-12

CONDITIONS: Correction of Nasolabial Folds

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Subdermal Injection — Injection of dermal filler
Device: Artiste Assisted Injection System — The Artiste™ Assisted Injection System is an air-powered device used to assist clinicians in injecting fluids into the body. The Artiste System was designed specifically to assist in the delivery of dermal fillers for the aesthetic correction of facial wrinkles, folds, and scars.

SUMMARY:
The purpose of this study is to characterize the safety and performance in normal therapeutic use of the Artiste System in comparison to standard manual administration of dermal fillers. Subjects are recruited from the investigator's practice and randomized to receive treatment with the Artiste System on either the left or right nasolabial fold, the contralateral fold to be treated with standard manual injections. Treatments occur in a single session to achieve optimal cosmetic results (OCR) balanced on both sides. Investigators are encouraged to use a variety of types and brands of dermal fillers, recruiting subjects for the study as necessary. Safety and performance evaluations will be made through a combination of clinical observations, questionnaires for the subject and for the Treating Investigator, and spontaneous reports of adverse events. There are 6 required study visits: Screening, Day 1 (Treatment Day), Day 3, Day 8, Day 15, and Day 29.

DETAILED DESCRIPTION:
This is a randomized, evaluator-blind, bilateral, controlled, multicenter study. Subjects are to be recruited from the investigator's practice and randomized to receive treatment with the Artiste System on either the left or right nasolabial fold, the contralateral fold to be treated with standard manual injections. Treatments will occur in a single session to achieve optimal cosmetic results (OCR) balanced on both sides. There are no specific requirements with respect to the type or brand of dermal filler to be used, but the investigators will be encouraged to use a variety of types and brands in the context of the study, recruiting subjects for the study as necessary. Safety and performance evaluations will be made through a combination of clinical observations (by a Blinded Evaluator distinct from the Treating Investigator), questionnaires for the subject and for the Treating Investigator, and spontaneous reports of adverse events. There will be a total of 6 required study visits: Screening, Day 1 (Treatment Day), Day 3, Day 8, Day 15, and Day 29.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age;
* Presenting at Screening with bilateral nasolabial folds rated 2 or greater on the Wrinkle Severity Rating Scale (SRS) by the Blinded Evaluator.
* Willing and able to provide informed consent;
* In good health, based upon the subject's report and medical history.

Exclusion Criteria:

* History of keloids, bleeding disorders, or severe allergic or anaphylactic reactions, including hypersensitivity to any components of the study materials;
* Active inflammatory process, scarring, or dense facial hair in the area of the nasolabial folds;
* Any chronic or acute medical condition that, in the opinion of the investigator, may interfere with evaluation of the study results or place the subject at undue risk;
* History of previous cosmetic treatment of the nasolabial folds within 6 months prior to the Screening visit;
* Planning to undergo facial surgery during the 4-week course of the study;
* Participation in a clinical investigation within the 30 days prior to the Screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Injection Site Reactions | 4 weeks
  Severity ratings.
Patient Acceptability | 4 weeks
  Questionnaire
Investigator Acceptability | 4 weeks
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Z. Paul Lorenc, MD, Principal Investigator — Independent
Locations (3):
- United States (3):
  - Z. Paul Lorenc, New York, New York
  - Suzanne Bruce & Associates, Houston, Texas
  - Premier Clinical Research, Spokane, Washington